CLINICAL TRIAL: NCT06834009
Title: A Phase 1, Open-label, Taste Assessment Study of Suzetrigine Spray-dried Dispersion in Healthy Adult Panelists
Brief Title: A Study of Suzetrigine (SUZ) Spray-dried Dispersion (SSD) in Healthy Adult Panelists
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VX24-548-020
Record Dates: First submitted 2025-02-13; First posted 2025-02-19 (Actual); Last update posted 2025-05-14 (Actual); Status verified 2025-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- SUZ (Experimental): Participants will be given SUZ SDD to retain in their mouths for approximately 10 seconds and then expectorate.
  Interventions: Drug: SUZ

INTERVENTIONS:
Drug: SUZ — Powder for oral administration.
  Other Names: VX-548

SUMMARY:
The purpose of this study is to evaluate the sensory attributes (basic tastes, aroma, texture, mouthfeel) of SUZ SDD and assess the impact of the dose on the sensory attributes.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4) (A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

- Panelists are qualified based on training and experience. They will be required to detect, identify, recognize, and accurately describe different taste elements and flavor combinations.

Key Exclusion Criteria:

* History of any illness or clinical condition that, in the opinion of the investigator, might confound the results of the study or pose an additional risk to the participant
* Sensitivity to SUZ
* Pregnant, nursing, or planning to become pregnant during the study

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-04-24 (Actual); Study Completion 2025-04-24 (Actual)

PRIMARY OUTCOMES:
Flavor Assessment Based on Flavor Profile Method of Descriptive Sensory Analysis per American Society for Testing and Material (ASTM) Approved Sensory Evaluation Method | Periodic Intervals up to 30 minutes post oral administration

CONTACTS AND LOCATIONS:
Locations (1):
- Senopsys, LLC, Woburn, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing